CLINICAL TRIAL: NCT01663857
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 1b/2 Study of LY2228820, a p38 MAPK Inhibitor, Plus Gemcitabine and Carboplatin Versus Gemcitabine and Carboplatin for Women With Platinum-Sensitive Ovarian Cancer
Brief Title: A Study LY2228820 for Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12517; I1D-MC-JIAE (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-08-08; First posted 2012-08-13 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — ralimetinib; Carboplatin; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase 1b (Cohort 1) LY2228820 200 milligrams (mg) (Experimental): Cohort 1: Cycles 1-6 (21 day cycles)- LY2228820 200 mg administered orally every 12 hours on days 1-10. Gemcitabine 1000 milligrams per square meter (mg/m^2) administered intravenously (IV) over 30 minutes on days 3 and 10. Carboplatin dose Area Under Curve (AUC) 4 (maximum dose 600 mg) administered IV over 30 minutes on day 3..
  Cohort 1: Cycles 7+ (28 day cycles)- LY2228820 300 mg administered orally every 12 hours on days 1-14.
  Interventions: Drug: LY2228820; Drug: Carboplatin; Drug: Gemcitabine
- Phase 1b (Cohort 2) LY2228820 300 mg (Experimental): Cohort 2: Cycles 1-6 (21 day cycles)- LY2228820 300 mg administered orally every 12 hours on days 1-10. Gemcitabine 1000 mg/m^2 administered IV over 30 minutes on days 3 and 10. Carboplatin dose Area Under Curve (AUC) 4 (maximum dose 600 mg) administered IV over 30 minutes on day 3.
  Cohort 2: Cycles 7+ (28 day cycles)- LY2228820 300 mg administered orally every 12 hours on days 1-14.
  Interventions: Drug: LY2228820; Drug: Carboplatin; Drug: Gemcitabine
- Phase 2 (Arm A) LY2228820 200 mg (Experimental): Arm A: Cycles 1-6 (21 day cycles)- LY2228820 200 mg administered orally every 12 hours on days 1-10. Gemcitabine 1000 mg/m^2 administered IV over 30 minutes on days 3 and 10. Carboplatin dose Area Under Curve (AUC) 4 (maximum dose 600 mg) administered IV over 30 minutes on day 3.
  Arm A: Cycles 7+ (28 day cycles)- LY2228820 300 mg administered orally every 12 hours on days 1-14.
  Interventions: Drug: LY2228820; Drug: Carboplatin; Drug: Gemcitabine
- Phase 2 (Arm B) Placebo (Placebo Comparator): Arm B: Cycles 1-6 (21 day cycles)- Placebo administered orally every 12 hours on days 1-10. Gemcitabine 1000 mg/m^2 administered IV over 30 minutes on days 3 and 10. Carboplatin dose Area Under Curve (AUC) 4 (maximum dose 600 mg) administered IV over 30 minutes on day 3.
  Arm B: Cycle 7+ (28 day cycles)- Placebo administered orally on days 1-14 to maintain blind.
  Interventions: Drug: Carboplatin; Drug: Placebo; Drug: Gemcitabine

INTERVENTIONS:
Drug: LY2228820 — Administered Orally
  Arms: Phase 1b (Cohort 1) LY2228820 200 milligrams (mg); Phase 1b (Cohort 2) LY2228820 300 mg; Phase 2 (Arm A) LY2228820 200 mg
Drug: Carboplatin — Administered IV
Drug: Placebo — Administered Orally
  Arms: Phase 2 (Arm B) Placebo
Drug: Gemcitabine — Administered IV
  Other Names: Gemzar; LY188011

SUMMARY:
A study for women with ovarian cancer that has returned at least 6 months after platinum-based chemotherapy.

DETAILED DESCRIPTION:
Phase 1b is unblinded and will have a small number of participants that will take LY2228820 plus gemcitabine and carboplatin to test the safety of the combination and determine a recommended dose for the Phase 2 portion.

Phase 2 will be blinded and all study participants will receive carboplatin and gemcitabine. Participants of one group will receive LY2228820, and the other group will receive placebo.

If the participant achieves at least stable disease, there is a maintenance phase following the first 6 cycles. The participant will take either LY2228820 or placebo. The participant will continue therapy until disease progression or other discontinuation criteria are fulfilled.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with ovarian, fallopian tube, or primary peritoneal cancer
* Have been treated one time with a platinum-based chemotherapy and your disease has come back at least six months after you completed treatment
* Are able to swallow tablets
* Have given written informed consent prior to any study procedures
* Have adequate blood counts, hepatic and renal function
* Have performance status equal to or less than 2 on Eastern Cooperative Oncology Group (ECOG) scale
* Have negative pregnancy test, and if participant is of child bearing potential must use birth control while on study and for three months after stopping study drug

Exclusion Criteria:

* Have been previously treated with Gemcitabine for ovarian, fallopian tube or primary peritoneal cancer
* Are currently enrolled or discontinued less than 14 days from another clinical trial
* Have a history of inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Have taken certain medications or had grapefruit juice within 7 days of initial dose of study drug, as levels of the study drug may be affected.
* Must not be pregnant or breastfeeding.
* Have malignancy or metastasis of the central nervous system
* Have borderline malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2012-07; Primary Completion 2017-05-25 (Actual); Study Completion 2018-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9am-5pm Eastern time *UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (29):
- United States (19):
  - St Josephs Hospital and Medical Center, Phoenix, Arizona
  - Arizona Oncology Associates, P.C., Tucson, Arizona
  - Sarasota Memorial Hospital, Sarasota, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Barnes Jewish Hospital, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - SMO Sarah Cannon Research Inst., Nashville, Tennessee
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Austin, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Bedford, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Fort Worth, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology - The Woodlands, The Woodlands, Texas
  - US Oncology, The Woodlands, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Northwest Cancer Specialists PC, Vancouver, Washington
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenslopes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parkville
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven, Belgium
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greifswald
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Vergote I, Heitz F, Buderath P, Powell M, Sehouli J, Lee CM, Hamilton A, Fiorica J, Moore KN, Teneriello M, Golden L, Zhang W, Pitou C, Bell R, Campbell R, Farrington DL, Bell-McGuinn K, Wenham RM. A randomized, double-blind, placebo-controlled phase 1b/2 study of ralimetinib, a p38 MAPK inhibitor, plus gemcitabine and carboplatin versus gemcitabine and carboplatin for women with recurrent platinum-sensitive ovarian cancer. Gynecol Oncol. 2020 Jan;156(1):23-31. doi: 10.1016/j.ygyno.2019.11.006. Epub 2019 Nov 29. PMID 31791552

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in Phase 1b are considered to have completed the study if they experience a dose-limiting toxicity or completed the Pharmacokinetic (PK) sampling set. Participants in Phase 2 are considered to have completed if they die due to any cause or who are alive and on study at conclusion, but are off treatment.
Groups:
- Phase 1b: Cohort 1: LY2228820 + Gemcitabine + Carboplatin: Cohort 1:LY2228820 200 milligrams (mg) administered orally every 12 hours (hr) on Days 1-10 of a 21-day cycle (Cycles 1-6).
  Gemcitabine 1000 mg per square meter (m2) administered intravenously (IV) over 30 minutes (min) on Days 3 and 10 of a 21-day cycle.
  Carboplatin area under the concentration curve (AUC) 4 (maximum dose 600mg) IV over 30 min. on Day 3 of a 21-day cycle.
  Cohort 1: LY2228820 300 mg orally every 12 hr. on Days 1-14 of a 28 day cycle (Cycles 7+).
- Phase 1b: Cohort 2: LY2228820 + Gemcitabine + Carboplatin: Cohort 2: LY2228820 300 mg administered orally every 12 hr. on Days 1-10 of a 21-day cycle.
  Gemcitabine 1000 mg/m2 IV over 30 min. on Days 3 and 10 of a 21-day cycle.
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3 of a 21-day cycle.
  Cohort 2: LY2228820 300 mg orally every 12 hr. on Days 1-14 of a 28 day cycle (Cycles 7+).
- Phase 2: Arm A: LY2228820 + Gemcitabine + Carboplatin: Arm A: LY2228820 200 mg orally every 12 hr. on Days 1-10 of a 21-day cycle.
  Gemcitabine 1000 mg/m2 IV over 30 min. on Days 3 and 10 of a 21-day cycle.
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3 of a 21-day cycle.
  Arm A: LY2228820 300 mg orally every 12 hr. on Days 1-14 of a 28 day cycle (Cycles 7+)
- Phase 2: Arm B: Placebo + Gemcitabine + Carboplatin: Arm B: Placebo orally every 12 hrs. on Days 1-10 of a 21-day cycle.
  Gemcitabine 1000 mg/m2 IV over 30 min. on Days 3 and 10 of a 21-day cycle.
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3 of a 21-day cycle.
  Arm B: Placebo orally every 12 hr. on Days 1-14 of a 28 day cycle (Cycles 7+)
Period: Overall Study
Arm/Group | Phase 1b: Cohort 1: LY2228820 + Gemcitabine + Carboplatin | Phase 1b: Cohort 2: LY2228820 + Gemcitabine + Carboplatin | Phase 2: Arm A: LY2228820 + Gemcitabine + Carboplatin | Phase 2: Arm B: Placebo + Gemcitabine + Carboplatin
Started | 6 | 2 | 58 | 52
Received at Least One Dose of Study Drug | 6 | 2 | 58 | 52
Completed | 6 | 1 | 48 | 48
Not Completed | 0 | 1 | 10 | 4
Not completed — Withdrew Consent to Study Participation | 0 | 1 | 7 | 3
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Phase 1b: Cohort 1: LY2228820 +Gemcitabine+Carboplatin: Cohort 1:LY2228820 200 milligrams (mg) administered orally every 12 hours (hr) on Days 1-10 of a 21-day cycle (Cycles 1-6).
  Gemcitabine 1000 mg per square meter (m2) administered intravenously (IV) over 30 minutes (min) on Days 3 and 10.
  Carboplatin area under the concentration curve administered intravenously (IV) over 30 minutes (AUC) 4 (maximum dose 600mg) IV over 30 min. on Day 3.
  Cohort 1: LY2228820 300 mg orally every 12 hr. on Days 1-10 of a 21-day cycle (Cycles 1-6).
- Phase 1b: Cohort 2: LY2228820 +Gemcitabine+Carboplatin: Cohort 2: LY2228820 300 mg administered orally every 12 hr. on Days 1-10 of a 21-day cycle (Cycles 1-6).
  Gemcitabine 1000 mg/m2 administered IV over 30 min on Days 3 and 10.
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3.
  Cohort 2:LY2228820 300 mg orally every 12 hr. on Days 1-14 of a 28-day cycle (Cycles 7+).
- Arm A: LY2228820 + Gemcitabine + Carboplatin: Arm A:LY2228820 200 mg orally every 12 hr. on Days 1-10 of a 21-day cycle (Cycles 1-6).
  Gemcitabine 1000 mg/m2 IV over 30 min. on Days 3 and 10.
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3.
  Arm A:LY2228820 300 mg orally every 12 hr. on Days 1-14 of a 28 day cycle (Cycles 7+).
- Arm B Placebo + Gemcitabine +Carboplatin: Arm B: Placebo orally every 12 hrs. on Days 1-10 of a 21-day cycle (Cycles 1-6).
  Gemcitabine 1000 mg/m2 IV over 30 min. on Days 3 and 10.
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3.
  Arm B: Placebo orally every 12 hr. on Days 1-14 of a 28 day cycle (Cycles 7+).
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Cohort 1: LY2228820 +Gemcitabine+Carboplatin | Phase 1b: Cohort 2: LY2228820 +Gemcitabine+Carboplatin | Arm A: LY2228820 + Gemcitabine + Carboplatin | Arm B Placebo + Gemcitabine +Carboplatin | Total
Number analyzed (Participants) | 6 | 2 | 58 | 52 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (6.8) | 65.0 (5.7) | 60.9 (10.4) | 62.2 (9.2) | 61.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 58 | 52 | 118
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 6 | 1 | 57 | 49 | 113
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 0 | 0 | 11 | 9 | 20
  United States | 5 | 2 | 30 | 25 | 62
  Australia | 0 | 0 | 4 | 6 | 10
  Germany | 1 | 0 | 13 | 12 | 26
Maintenance Therapy as a Part of or After a First Line Platinum Regimen [Count of Participants; unit: Participants] — Population: Maintenance therapy as part of or after first line platinum regimen data was used as a cofactor in the analysis of Progression Free Survival (PFS). Zero participants analyzed for Phase 1 portion of the study.Data was collected only from participants treated in the Phase 2 portion of the study.
  Participants
    Received Maintenance Therapy: number analyzed (Participants) | 0 | 0 | 58 | 52 | 110
    Received Maintenance Therapy |  |  | 7 | 7 | 14
    Did Not Receive Maintenance Therapy: number analyzed (Participants) | 0 | 0 | 58 | 52 | 110
    Did Not Receive Maintenance Therapy |  |  | 15 | 15 | 30
    Data Missing or Not Collected: number analyzed (Participants) | 0 | 0 | 58 | 52 | 110
    Data Missing or Not Collected |  |  | 36 | 30 | 66

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Recommended Phase 2 Dose of LY2228820 in Combination With Gemcitabine and Carboplatin (Maximum Tolerated Dose [MTD])
Description: Recommended Phase 2 dose of LY2228820 that could be safely administered in combination with gemcitabine and carboplatin based on defined dose limiting toxicities (DLT) assessment and MTD definition. The MTD is defined as the highest dose level at which no more than 33% of patients experience a DLT during Cycle 1 that does not exceed the single-agent MTD for LY2228820 (300 mg Q12H).
Time Frame: Cycle 1 (21 Days)
Population: All participants who received at least one dose of study drug in Phase 1b.
Measure: Number; unit: milligrams (mg)
Groups:
- LY2228820 + Gemcitabine + Carboplatin: Cohort 1 : LY2228820 200 milligrams (mg) administered orally every 12 hours (hr) on Days 1-10 of a 21-day cycle (Cycles 1-6)
  Gemcitabine 1000 mg per square meter (m2) administered intravenously (IV) over 30 minutes (min) on Days 3 and 10
  Carboplatin area under the concentration curve (AUC) 4 (maximum dose 600mg) IV over 30 min. on Day 3
  Cohort 2: LY2228820 300 mg administered orally every 12 hr. on Days 1-10
  Gemcitabine 1000 mg/m2 IV over 30 min. on Days 3 and 10
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3
  Cohort 1 and 2: LY2228820 300 mg orally every 12 hr. on Days 1-14 of a 28 day cycle (Cycles 7+)
Arm/Group | LY2228820 + Gemcitabine + Carboplatin
Number analyzed (Participants) | 8
milligrams (mg) | 200

2. Primary Outcome: Phase 2: Progression-free Survival (PFS) in Participants Treated With LY2228820 Plus Gemcitabine and Carboplatin Versus Placebo Plus Gemcitabine and Carboplatin
Description: PFS was defined as time from date of randomization to the date of investigator-determined objective progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death due to any cause, whichever occurred first. Progressive disease (PD) is defined as at least a 20% increase in the sum of the largest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Randomization to Date of Disease Progression or Death from any cause (up to 3 years)
Population: All participants in Phase 2 who received at least one dose of study drug.
Measure: Median (90% Confidence Interval); unit: months
Groups:
- LY2228820 + Gemcitabine +Carboplatin: Arm A: LY2228820 200 mg orally every 12 hr. on Days 1-10 of 21-day cycles.
  Gemcitabine 1000 mg/m2 IV over 30 min on Days 3 and 10 of 21-day cycles.
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3 of 21-day cycles.
  Arm A: LY2228820 300 mg orally every 12 hr. on Days 1-14 of a 28-day cycle (Cycles 7+)
- Placebo + Gemcitabine + Carboplatin: Arm B: Placebo orally every 12 hrs. on Days 1-10 of 21-day cycles.
  Gemcitabine 1000 mg/m2 IV over 30 min on Days 3 and 10 of 21-day cycles.
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. n Day 3 of 21-day cycles.
  Arm B: Placebo orally every 12 hr. on Days 1-14 of a 28-day cycle (Cycles 7+)
Arm/Group | LY2228820 + Gemcitabine +Carboplatin | Placebo + Gemcitabine + Carboplatin
Number analyzed (Participants) | 58 | 52
months | 10.25 [7.85 to 10.87] | 8.44 [7.56 to 9.33]
Statistical Analysis 1: Comparison: LY2228820 + Gemcitabine +Carboplatin vs Placebo + Gemcitabine + Carboplatin; Test type: Superiority; p = 0.4, Log Rank

3. Secondary Outcome: Phase 2: Percentage of Participants Who Achieve Complete Response or Partial Response (Overall Response Rate)
Description: Overall Response Rate was estimated as the percentage of participants with best response of Complete Response (CR) or Partial Response (PR), based on RECIST version 1.1 divided by the total number of randomized participants. CR is defined as disappearance of all target lesions. PR is defined as at least 30% disease in the sum of the largest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Baseline to Disease Progression (up to 3 years)
Population: All participants who received at least one dose of study drug in Phase 2.
Measure: Number; unit: percentage of participants
Groups:
- LY2228820 + Gemcitabine +Carboplatin: Arm A: LY2228820 200 mg orally every 12 hr. on Days 1-10 of a 21-day cycle.
  Gemcitabine 1000 mg/m2 IV over 30 min.(+ 15 min.) on Days 3 and 10 of a 21-day cycle.
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3 of a 21-day.
  Arm A: LY2228820 300 mg orally every 12 hr. on Days 1-14 of a 28-day cycle (Cycles 7+).
- Placebo + Gemcitabine + Carboplatin: Arm B: Placebo orally every 12 hrs. on Days 1-10 of a 21-day cycle.
  Gemcitabine 1000 mg/m2 IV over 30 min. on Days 3 and 10 of a 21-day cycle.
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3 of a 21-day cycle.
  Arm B: Placebo orally every 12 hr. on Days 1-14 of a 28-day cycle (Cycles 7+)
Arm/Group | LY2228820 + Gemcitabine +Carboplatin | Placebo + Gemcitabine + Carboplatin
Number analyzed (Participants) | 58 | 52
percentage of participants | 46.6 | 46.2

4. Secondary Outcome: Phase 2: Overall Survival
Description: Data presented are the median overall survival in months for participants in the Phase 2 treatment arms.
Time Frame: Baseline to Date of Death from any cause (up to 5 years)
Population: All participants in Phase 2 who received at least one dose of drug.
Measure: Median (90% Confidence Interval); unit: months
Groups:
- LY2228820 + Gemcitabine +Carboplatin: Arm A: LY2228820 200 mg orally every 12 hr. on Days 1-10 of a 21-day cycle.
  Gemcitabine 1000 mg/m2 IV over 30 min. on Days 3 and 10 of a 21-day cycle.
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3 of a 21-day.
  Arm A: LY2228820 300 mg orally every 12 hr. on Days 1-14 of a 28-day cycle (Cycles 7+).
Arm/Group | LY2228820 + Gemcitabine +Carboplatin | Placebo + Gemcitabine + Carboplatin
Number analyzed (Participants) | 58 | 52
months | 29.17 [23.26 to 52.40] | 25.10 [21.95 to 33.68]
Statistical Analysis 1: Comparison: LY2228820 + Gemcitabine +Carboplatin vs Placebo + Gemcitabine + Carboplatin; Test type: Superiority; p = 0.4686, Log Rank

5. Secondary Outcome: Phase 1b and 2: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to 8 Hours (AUC 0-8) of LY2228820
Description: PK parameters after administration of LY2228820 for both Phase 1b and Phase 2.
Time Frame: Phase1b:Cycle(C)1 Day(D)1:Predose(PRD),0.5,1,2,4,6,8 hours(hr)postdose(PD); C1D10:PRD,0.5,1,2,8hrPD; C2D10:PRD,0.5,1,2,4,6,8,12hrPD; C7D3:PRD,0.5,1,2,4,6hrPD; Phase 2: C1D3:PRD,0.5,1,2,4,6,8hrPD; C1D10:PRD,0.5,1,2,4,6,8hrPD; C7D3:PRD,0.5,1,2,4,6,8hrPD
Population: All participants in Phase 1b and Phase 2 who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms * hr per milliliter (ng*hr/mL)
Groups:
- 200 mg LY2228820: Phase 1b (Cohort 1) and Phase 2 (Arm A): LY2228820 200 mg administered orally every 12 hours on Days 1-10, Cycles 1-6 of a 21 day cycle.
  .
- 300 mg LY2228820: Phase 1b (Cohort 2) and Phase 2 (Arm A) in the maintenance portion with LY2228820 300 mg administered orally every 12 hours on Days 1-14 Cycle 7+ of a 28-day cycle.
Arm/Group | 200 mg LY2228820 | 300 mg LY2228820
Number analyzed (Participants) | 13 | 10
nanograms * hr per milliliter (ng*hr/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 2
  Cycle 1 Day 1 | 3470 (91) | 3560 (1)
  Cycle 1 Day 3: number analyzed (Participants) | 7 | 0
  Cycle 1 Day 3 | 3170 (22) |
  Cycle 1 Day 10: number analyzed (Participants) | 11 | 1
  Cycle 1 Day 10 | 4270 (62) | 9350 (NA) — Due to n of 1 individual value provided.
  Cycle 2 Day 10: number analyzed (Participants) | 5 | 1
  Cycle 2 Day 10 | 3270 (38) | 3490 (NA) — Due to n of 1 individual value provided.
  Cycle 7 Day 3: number analyzed (Participants) | 0 | 10
  Cycle 7 Day 3 |  | 7230 (72)

6. Secondary Outcome: Phase 2: Change From Baseline in Functional Assessment of Cancer Therapy-Ovarian Cancer (FACT-O) Total Score
Description: The Functional Assessment of Cancer Therapy-Ovarian Cancer (FACT-O) instrument measures health related quality of life (HRQoL) in participants with ovarian cancer. The instrument is organized into sections of physical, social/family, emotional, functional well-being and ovarian subscales with a 5-point rating scale in which 0 = "not at all" and 4 = "very much." Data presented here are change from baseline at follow-up in the FACT-O Total Score. The total score is the sum of Physical Well Being (PWB) + Social Well-being (SWB) + Emotional Well Being (EWB) + Family Well-being (FWB) + Ovarian Cancer Subscale (OCS). The FACT-O Total score range 0 - 152 with higher scores indicating better quality of life.
Time Frame: Baseline, Study Completion (up to 3 years)
Population: All participants in Phase 2 who received at least one dose of study drug and had at least one post baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- LY2228820 + Gemcitabine +Carboplatin: Arm A: LY2228820 200 mg orally every 12 hr. on Days 1-10 of a 21-day cycle.
  Gemcitabine 1000 mg/m2 IV over 30 min. on Days 3 and 10 of a 21-day cycle.
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3 of a 21-day.
  Arm A: LY2228820 300 mg orally every 12 hr. on Days 1-14 of a 28 day cycle (Cycles 7+)
- Placebo + Gemcitabine + Carboplatin: Arm B: Placebo orally every 12 hrs. on Days 1-10 of a 21-day cycle.
  Gemcitabine 1000 mg/m2 IV over 30 min. on Days 3 and 10 of a 21-day cycle.
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3 of a 21-day cycle.
  Arm B: Placebo orally every 12 hr. on Days 1-14 of a 28 day cycle (Cycles 7+)
Arm/Group | LY2228820 + Gemcitabine +Carboplatin | Placebo + Gemcitabine + Carboplatin
Number analyzed (Participants) | 58 | 52
units on a scale | -0.6 (21.14) | -8.9 (19.92)

ADVERSE EVENTS:
Time Frame: Up to 4.5 years
Description: All participants who received at least one dose of drug.
Groups:
- Phase 1b: Cohort 1: LY2228820 + Gemcitabine + Carboplatin: Cohort 1: LY2228820 200 milligrams (mg) administered orally every 12 hours (hr) on Days 1-10 of a 21-day cycle (Cycles 1-6)
  Gemcitabine 1000 mg per square meter (m2) administered intravenously (IV) over 30 minutes (min) on Days 3 and 10
  Carboplatin area under the concentration curve (AUC) 4 (maximum dose 600mg) IV over 30 min. on Day 3
  Cohort 1: LY2228820 300 mg orally every 12 hr. on Days 1-14 of a 28 day cycle (Cycles 7+)
- Phase 1b: Cohort 2: LY2228820 + Gemcitabine + Carboplatin: Cohort 2: LY2228820 300 mg administered orally every 12 hr. on Days 1-10
  Gemcitabine 1000 mg/m2 IV over 30 min. on Days 3 and 10
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3
  Cohort 2: LY2228820 300 mg orally every 12 hr. on Days 1-14 of a 28 day cycle (Cycles 7+)
- Phase 2: Arm A: LY2228820 + Gemcitabine + Carboplatin: Arm A: LY2228820 200 mg orally every 12 hr. on Days 1-10
  Gemcitabine 1000 mg/m2 IV over 30 min. on Days 3 and 10
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3
  Arm A: LY2228820 300 mg orally every 12 hr. on Days 1-14 of a 28 day cycle (Cycles 7+)
- Phase 2: Arm B: Placebo + Gemcitabine + Carboplatin: Arm B: Placebo orally every 12 hrs. on Days 1-10
  Gemcitabine 1000 mg/m2 IV over 30 min. on Days 3 and 10
  Carboplatin AUC 4 (maximum dose 600mg) IV over 30 min. on Day 3
  Arm B: Placebo orally every 12 hr. on Days 1-14 of a 28 day cycle (Cycles 7+)
Arm/Group | Phase 1b: Cohort 1: LY2228820 + Gemcitabine + Carboplatin | Phase 1b: Cohort 2: LY2228820 + Gemcitabine + Carboplatin | Phase 2: Arm A: LY2228820 + Gemcitabine + Carboplatin | Phase 2: Arm B: Placebo + Gemcitabine + Carboplatin
All-Cause Mortality (participants affected / at risk) | 3/6 | 1/2 | 30/58 | 31/52
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/2 | 26/58 | 12/52
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2 | 58/58 | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Cohort 1: LY2228820 + Gemcitabine + Carboplatin (N=6) | Phase 1b: Cohort 2: LY2228820 + Gemcitabine + Carboplatin (N=2) | Phase 2: Arm A: LY2228820 + Gemcitabine + Carboplatin (N=58) | Phase 2: Arm B: Placebo + Gemcitabine + Carboplatin (N=52)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (7) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (5) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (3) | 0 (0) | 2 (2) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (6) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Pelvic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urostomy complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nuclear magnetic resonance imaging abdominal abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Cohort 1: LY2228820 + Gemcitabine + Carboplatin (N=6) | Phase 1b: Cohort 2: LY2228820 + Gemcitabine + Carboplatin (N=2) | Phase 2: Arm A: LY2228820 + Gemcitabine + Carboplatin (N=58) | Phase 2: Arm B: Placebo + Gemcitabine + Carboplatin (N=52)
Anaemia (Blood and lymphatic system disorders) | 5 (8) | 1 (4) | 32 (91) | 25 (73)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (8) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 5 (24) | 2 (4) | 26 (72) | 26 (74)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (9) | 0 (0) | 17 (40) | 14 (47)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 6 (6) | 8 (9)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (4)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (6) | 12 (13)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 12 (13) | 8 (9)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 5 (7)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (5) | 1 (1) | 23 (31) | 22 (24)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 1 (1) | 23 (40) | 14 (18)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Nausea (Gastrointestinal disorders) | 4 (8) | 0 (0) | 31 (39) | 33 (50)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 9 (10) | 10 (11)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 17 (23) | 12 (12)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Fatigue (General disorders) | 5 (11) | 0 (0) | 40 (50) | 38 (48)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 7 (9) | 7 (8)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 8 (9) | 6 (7)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 5 (7) | 5 (5)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 3 (3)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 3 (4) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (6) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 8 (14) | 7 (10)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 7 (8) | 6 (11)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (5) | 1 (2) | 25 (42) | 13 (35)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 0 (0) | 17 (28) | 10 (22)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 9 (12) | 7 (7)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 3 (5)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 26 (76) | 29 (92)
Platelet count decreased (Investigations) | 1 (6) | 1 (2) | 21 (53) | 20 (66)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 3 (5)
White blood cell count decreased (Investigations) | 3 (12) | 0 (0) | 20 (47) | 19 (55)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 14 (15) | 12 (13)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (4) | 3 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (5) | 4 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 7 (11) | 5 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (6) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 7 (10) | 12 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (7) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 12 (13) | 9 (9)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5) | 5 (5)
Headache (Nervous system disorders) | 3 (4) | 0 (0) | 10 (10) | 12 (20)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (3) | 0 (0) | 5 (6) | 2 (2)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 6 (7) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 4 (5) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 3 (3) | 4 (4)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 11 (11) | 12 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 17 (20) | 9 (10)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 5 (6) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 7 (7) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 7 (7) | 3 (3)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 10 (10) | 10 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 7 (10) | 5 (7)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (5) | 3 (6)
Social problem (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT01663857/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT01663857/SAP_001.pdf